CLINICAL TRIAL: NCT07302009
Title: Safety and Efficacy of Bladder Temperature Monitoring-Guided Targeted Temperature Management in Patients With Severe : A Multicenter Randomized Controlled Trial
Brief Title: Targeted Temperature Management Via Bladder Monitoring in ICH
Acronym: BTTM-ICH
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Yanyan Gong (Other)
Collaborators: First Affiliated Hospital of Gannan Medical University (Other); Xiangya Hospital of Central South University (Other); Renmin Hospital of Wuhan University (Other); Zhejiang University (Other); The First People's Hospital of Changde City (Other); The First People's Hospital of Xiushui (Other); Yichang Central People's Hospital (Other)
Responsible Party: Sponsor-Investigator, Yanyan Gong, Senior Nurse, Department of Neurosurgery, The Second Affiliated Hospital of Nanchang University, Second Affiliated Hospital of Nanchang University
Organization: Second Affiliated Hospital of Nanchang University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: IIT-I-2025-093
Record Dates: First submitted 2025-12-11; First posted 2025-12-24 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-12

CONDITIONS: Intracerebral Hemorrhage; Targeted Temperature Management
Keywords: Intracerebral Hemorrhage; Targeted Temperature Management; Bladder Temperature Monitoring
MeSH Terms: conditions — Cerebral Hemorrhage

STUDY DESIGN:
Intervention Model Description: Only the outcome assessors and the statistical analysis team will be masked to group allocation. The treating clinicians and patients are unmasked.
Who Masked: Outcomes Assessor
Masking Description: Only the outcome assessors and the statistical analysis team will be masked to group allocation. The treating clinicians and patients are unmasked.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Bladder Temperature Monitoring Group (Experimental): Patients in this arm will receive Targeted Temperature Management (TTM) guided by continuous, real-time core temperature monitoring via a bladder thermometer. TTM may include therapeutic hypothermia (TH, 32.0°C ≤ temp < 36.0°C), normothermia control (36.0-37.5°C), or fever treatment, as clinically indicated. Temperature is recorded hourly.
  Interventions: Device: Bladder Temperature Monitoring
- Standard Temperature Monitoring Group (Active Comparator): Patients in the control arm will receive Targeted Temperature Management (TTM) guided by intermittent axillary temperature measurements using a mercury-in-glass thermometer, recorded every four hours. TTM may include therapeutic hypothermia, maintenance of normothermia, or treatment of fever, as clinically indicated.
  Interventions: Device: Standard Temperature Monitoring Group

INTERVENTIONS:
Device: Bladder Temperature Monitoring — This intervention utilizes a single-use, sterile, thermometric silicone urinary catheter that, upon insertion, provides continuous, real-time measurement of core body temperature, which is used to dynamically guide all phases of Targeted Temperature Management (TTM).
  Arms: Bladder Temperature Monitoring Group
Device: Standard Temperature Monitoring Group — Axillary temperature is measured intermittently using a mercury-in-glass thermometer. The thermometer is placed in the axilla for a standardized period (e.g., 5-10 minutes) to obtain a reading. Temperature data is recorded every 4 hours and is used to guide adjustments in Targeted Temperature Management (TTM) therapy.
  Arms: Standard Temperature Monitoring Group

SUMMARY:
The goal of this clinical trial is to learn whether a bladder temperature monitoring-guided targeted temperature management (TTM) strategy improves functional recovery in patients with severe intracerebral hemorrhage, compared to conventional temperature monitoring. It will also assess the safety of this monitoring approach. The main questions it aims to answer are:

* Does continuous bladder temperature monitoring-guided TTM improve the likelihood of a favorable functional outcome (modified Rankin Scale score 0-2) at 180 days after onset?
* What medical problems (such as infections, shivering, deep vein thrombosis, or sepsis) do participants experience while under the TTM strategy? Researchers will compare the intervention group (using continuous bladder temperature monitoring) with the control group (using conventional intermittent temperature monitoring with a mercury thermometer at the armpit) to see if the bladder temperature-guided TTM strategy leads to better outcomes.

Participants will:

* Be randomly assigned to one of the two temperature monitoring strategies
* Receive standard medical and surgical care for severe intracerebral hemorrhage

DETAILED DESCRIPTION:
Neurogenic fever, a non-infectious febrile condition, is relatively common following severe brain injuries such as intracerebral hemorrhage, aneurysmal subarachnoid hemorrhage, and acute ischemic stroke. Early-onset fever may represent a systemic response to the brain injury itself, whereas late-onset fever is often attributable to severe stroke complications, including infection and deep vein thrombosis (DVT). Fever is positively correlated with illness severity. Substantial evidence confirms that hyperthermia significantly increases the risk of complications-such as rebleeding, exacerbated cerebral edema, seizures-and mortality in patients with intracerebral hemorrhage, and is associated with poor prognosis. Studies have found that mortality and voluntary discharge rates in stroke patients with extreme hyperthermia are six times higher than those in patients with normal body temperature. This underscores the critical importance of timely and effective temperature control and management in stroke patients, which has been shown to reduce mortality and improve neurological outcomes.

Body temperature is a vital sign and a key indicator of health status. Under the regulation of the hypothalamic thermoregulatory center, it fluctuates within a narrow range; deviations beyond this range suggest potential abnormalities [8]. In severe ICH patients, temperature fluctuations not only reflect systemic stress but also serve as a sensitive indicator of intracranial pathological changes, such as hematoma expansion, progressing cerebral edema, and secondary brain injury. However, a critical issue in current clinical practice is the frequent failure to detect temperature changes in severe ICH patients promptly. Typically, significant temperature elevations or reductions are only recognized when they reach extreme levels. This makes it exceptionally difficult to identify the onset of temperature changes, the timing of peaks/troughs, and the effective time of interventions, severely hindering the early recognition of clinical deterioration and timely intervention, potentially missing critical windows for improving outcomes. Therefore, continuous temperature monitoring is crucial for severe ICH patients, particularly given their high fever incidence and elevated risk of secondary brain injury; fever must be identified and managed aggressively upon onset.

Intracranial temperature (ICT) can be measured via direct (e.g., intraparenchymal, intraventricular, subdural catheters) or indirect methods. However, direct measurement is invasive, its application is limited in ICH patients with coagulopathies or high rebleeding risks, and it carries additional risks of hemorrhage or infection. When direct ICT monitoring probes or devices are unavailable, it is recommended to use core temperature measurements from sites that closely approximate and are relatively stable compared to brain temperature. Core temperature measurement sites include the tympanic membrane, temporal artery, rectum, bladder, esophagus, and pulmonary artery. The temperature monitored via a pulmonary artery catheter is considered closest to the true core temperature. Expert consensus on targeted temperature management (TTM) in neurocritical care recommends a preference for brain temperature measurement, followed by esophageal and bladder temperatures. However, esophageal temperature measurement is mildly invasive. Although bladder temperature is recommended by consensus and is known to reliably reflect core temperature trends, in-depth research and direct evidence regarding its application specifically in the high-risk ICH population, particularly rigorous comparative data against the gold standard of intracranial temperature, remain notably scarce.

Given the high fever rate in severe ICH patients, the decisive impact of temperature management on prognosis, the limitations of existing core temperature monitoring methods (especially esophageal) in this population, and the lack of high-quality evidence for bladder temperature monitoring, exploring an accurate, reliable, and practical method for continuous core temperature monitoring suitable for severe ICH patients is of urgent clinical significance. Bladder temperature monitoring offers significant advantages: its readings closely approximate intracranial core temperature trends, enabling real-time reflection of patient temperature fluctuations; it boasts high measurement accuracy and relatively simple operation; it can be implemented via the indwelling urinary catheter routinely placed in severe ICH patients (for monitoring urine output and managing retention), without adding significant nursing workload, avoiding additional invasive procedures, and minimizing patient disturbance, sleep disruption, and treatment interference, while allowing for stable, prolonged placement. More importantly, the continuous monitoring capability of bladder temperature can empower clinicians to grasp the dynamic temperature changes in severe ICH patients in real-time, providing crucial information for the early detection of fever and potential clinical deterioration (e.g., infection, hematoma expansion, worsening cerebral edema), thereby securing a valuable early intervention time window for implementing neuroprotective strategies and complication prevention.

In recent years, bladder temperature monitoring has gained attention in temperature management due to its relative operational simplicity, close approximation to core temperature, and suitability for continuous monitoring. However, current research on using bladder temperature monitoring to guide TTM in neurocritical care patients, specifically those with spontaneous intracerebral hemorrhage, is relatively limited. Existing studies often focus on investigating the impact of TTM itself on patient outcomes or validating the correlation between bladder temperature and traditional monitoring techniques. The updated consensus guidelines from the Neuroprotective Therapy Consensus Review Group emphasize that core temperature is the most important surrogate for intracranial temperature and note that implementing TTM requires reliance on technology capable of real-time, continuous temperature monitoring to precisely regulate body temperature and adjust treatment strategies promptly.

Therefore, this study aims to conduct a randomized controlled trial directly comparing the safety and efficacy of bladder temperature monitoring-guided TTM (intervention group) versus conventional temperature monitoring (axillary temperature)-guided management (control group) in severe ICH patients. The primary efficacy endpoint will assess neurological outcome. Through this research, we seek to evaluate its value in improving key clinical outcomes (neurological recovery) and ensuring patient safety, thereby guiding clinical practice, improving prognosis, and providing new evidence-based medical evidence.

ELIGIBILITY:
Inclusion Criteria:

1. Neurocritical care patients: Study subjects are patients with first-time spontaneous intracerebral hemorrhage.
2. Age ≥ 18 years and ≤ 85 years.
3. Glasgow Coma Scale (GCS) score ≤ 8 at ICU admission.
4. For supratentorial ICH: Hematoma volume < 60 mL. For subarachnoid hemorrhage (SAH): Modified Fisher grade ≥ 2, and the aneurysm has been treated with endovascular intervention.
5. Pre-morbid modified Rankin Scale (mRS) score of 0 or 1.
6. Signed informed consent provided by a legally authorized representative.

Exclusion Criteria:

1. Fever (≥38.0°C) that lasted over 1 hour or occurred more than once prior to enrollment.
2. Pre-existing neurological, psychiatric, or other comorbidities that may compromise the assessment of neurological or functional outcomes.
3. Underlying conditions with a life expectancy of less than 6 months, estimated prior to onset.
4. Severe injury indicative of poor prognosis: brain death, receiving palliative care only, or irreversible brain injury.
5. Pregnancy.
6. Unilateral or bilateral pupillary dilation.
7. Currently participating in other investigational/interventional clinical trials (involving medical devices or drugs).
8. Subjects deemed ineligible for enrollment by the investigator.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 308 (Estimated)
Dates: Start 2026-01-20 (Estimated); Primary Completion 2027-12-30 (Estimated); Study Completion 2027-12-30 (Estimated)

PRIMARY OUTCOMES:
Percentage of patients with mRS 0-2 at 180 days post-onset | 180 days post-onset（±14 days）
  The proportion of participants achieving a favorable functional outcome, defined as a modified Rankin Scale (mRS) score of 0 to 2, at 180 days (±14 days) post-onset. The mRS is a standardized measure of neurological disability ranging from 0 (no symptoms) to 6 (death). A score of 0-2 represents a favorable functional outcome.

SECONDARY OUTCOMES:
Daily mean fever burden | From enrollment until ICU discharge, meeting hospital discharge criteria, or up to 14 days (336 hours) (whichever occurs first)
  Calculated as the area under the curve (AUC) of temperature above the fever threshold (defined as ≥38.0°C)
Total hospitalization costs | From enrollment until hospital discharge
Percentage of patients with mRS 0-2 at 90 days post-onset. | 90 days post-onset（±14 days）
Neurological function assessed by GOS at 90 days | 90 days post-onset（±14 days）
Neurological function assessed by NIHSS at 90 days | 90 days post-onset（±14 days）
Neurological function assessed by GOS at 180 days | 180 days post-onset（±14 days）
Neurological function assessed by NIHSS at 180 days | 180 days post-onset（±14 days）
Barthel Index scores at 90 and 180 days after onset. | 90 (±14 days) and 180 (±14 days) days post-onset
Length of stay in the Intensive Care Unit (ICU) | From ICU admission until ICU discharge
Total duration of hospital stay | From enrollment until hospital discharge
Infection rate (pneumonia, urinary tract infection) | From ICU admission until ICU discharge
DVT Incidence | From ICU admission until ICU discharge
Sepsis Incidence | From ICU admission until ICU discharge
Malignant Edema Incidence | From ICU admission until ICU discharge
All-cause mortality | All-cause mortality within 180 days post onset

IPD SHARING:
Plan to Share IPD: No